CLINICAL TRIAL: NCT04665453
Title: Comparison of Efficacy of Dexmedetomidine and Melatonin for Sleep Induction for Electroencephalography in Children
Brief Title: Dexmedetomidine and Melatonin for Sleep Induction for EEG in Children
Acronym: MeloDex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Damjan Osredkar, Assoc. Prof. Damjan Osredkar, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0120-597/2019/16
Record Dates: First submitted 2020-12-02; First posted 2020-12-11 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Electroencephalography; Child; Dexmedetomidine; Melatonin; Sleep; Epilepsy
Keywords: Child; Dexmedetomidine; Melatonin; Electroencephalography; Autism Spectrum Disorder; Developmental Delay Disorder; Epilepsy; Sleep; Sleep induction
MeSH Terms: conditions — Epilepsy; Autism Spectrum Disorder; Developmental Disabilities | interventions — Electroencephalography; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Melatonin peroral (Experimental): 0,1mg/kg melatonin will be given in the form of a syrup to the participant before EEG and vital functions monitoring
  Interventions: Diagnostic Test: Electroencephalography; Diagnostic Test: Monitoring of vital functions; Drug: Melatonin 0,1mg/kg oral syrup
- Dexmedetomidine intranasally (Experimental): 3 mcg/kg of dexmedetomidine in the form of a nasal spray will be given to the participant before EEG and vital functions monitoring
  Interventions: Diagnostic Test: Electroencephalography; Diagnostic Test: Monitoring of vital functions; Drug: Dexmedetomidine 3 mcg/kg intranasally
- Dexmedetomidine sublingually (Experimental): 3 mcg/kg of dexmedetomidine will be given to the participant sublingually before EEG and vital functions monitoring
  Interventions: Diagnostic Test: Electroencephalography; Diagnostic Test: Monitoring of vital functions; Drug: Dexmedetomidine 3 mcg/kg sublingually

INTERVENTIONS:
Diagnostic Test: Electroencephalography — Recording of the brain electrical activity during sleep; background activity and sleep phases will be evaluated
  Other Names: EEG
Diagnostic Test: Monitoring of vital functions — Measuring of respiratory rate, heart rate, SpO2, every 10 minutes after the medicine is given to the patient for the duration of EEG, and after 120 minutes. Blood pressure is measured at the time of application of the medicine, at the end of EEG and after 120 minutes.
Drug: Melatonin 0,1mg/kg oral syrup — Melatonine in the form of syrup will be given orally to child.
  Arms: Melatonin peroral
Drug: Dexmedetomidine 3 mcg/kg sublingually — Dexmedetomidine in the form of a solution will be given to child sublingually.
  Arms: Dexmedetomidine sublingually
Drug: Dexmedetomidine 3 mcg/kg intranasally — Dexmedetomidine in the form of nasal spray will be given to child intranasally.
  Arms: Dexmedetomidine intranasally

SUMMARY:
The aim of the study is to compare the effect of melatonin, given orally, dexmedetomidine, given intranasally, and dexmedetomidine given sublingually on sleep induction, sleep duration, their possible impact on vital functions and technical implementation of EEG.

DETAILED DESCRIPTION:
At University Medical Centre Ljubljana (UMCL; Slovenia), the investigators use electroencephalography (EEG) in wakefulness and sleep for diagnostic and therapeutic purposes in children with (suspected) epilepsy. Since epileptiform activity can only be detected during sleep in some patients and because children with intellectual disabilities have sometimes problems with cooperation, EEG in induced sleep is required.

In this study, the investigators will enroll 150 children who need EEG recorded in their sleep. The investigators will compare safety and efficacy of the two active substances, one of which will be given in two possible routes. Fifty children will receive melatonin in the form of a syrup orally, 50 children will receive dexmedetomidine intranasally in the form of a nasal spray, and 50 children will receive dexmedetomidine sublingually. The investigators will monitor the following parameters: the time in which the child falls asleep, vital functions during sleep (blood pressure, blood oxygen saturation, respiratory rate frequency and heart rate frequency), the impact on the technical implementation of EEG, the depth of sleep and waking time. All parents will give their written consent for their child to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 20 years
* Referral for EEG in sleep
* Children/young adults whose parents/caregivers were informed about the aims of the study and have signed the Informed consent form

Exclusion Criteria:

* Children that were unable to follow the study protocol were excluded during the study

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the three medical interventions on sleep initiation | During the intervention
  The time-interval between the drug application and time of sleep initiation will be recorded in minutes. These values will be compared across the three arms of the study
Comparison of the three medical interventions on the depth of sleep and the most prominent sleep stage on EEG | During the intervention
  During EEG in sleep, which will be recorderd using a standard 10-20 placement with additional electrodes for breathing and ECG, the EEG background activity will be evaluated for the deepest sleep stage according to the standard EEG classification (Carskadon MA, Dement WC. Normal Human Sleep: an Overview. In: Kryger M, Roth T, Dement WC. Principles and practice of sleep medicine. St.Louis: Saunders/Elsevier, 2011:16-26.). Also, the sleep stage in which the patient will spend the most time will be noted. These values will be compared across the three arms of the study.

SECONDARY OUTCOMES:
Comparison of the three medical interventions on respiratory rate | During the intervention
  Measurement of respiratory rate every 10 minutes after the medicine is given to the patient for the duration of EEG recording, and after 120 minutes. The values will be compared across the three arms of the study.
Comparison of the three medical interventions on heart rate | During the intervention
  Measurement of heart rate every 10 minutes after the medicine is given to the patient for the duration of EEG recording, and after 120 minutes. The values will be compared across the three arms of the study.
Comparison of the three medical interventions on oxygene saturation | During the intervention
  Measurement of oxygene saturation using pulse oximetry every 10 minutes after the medicine is given to the patient for the duration of EEG recording, and after 120 minutes. The values will be compared across the three arms of the study.
Comparison of the three medical interventions on blood pressure | During the intervention
  Measurement of systolic and diastolic blood pressure will be noted at the time of application of the medicine, at the end of EEG and after 120 minutes. These values will be compared across the three arms of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peganc Nuncic K, Neubauer D, Orazem Mrak J, Perkovic Benedik M, Mahne U, Bizjak N, Rener Primec Z, Sustar N, Butenko T, Vrscaj E, Osredkar D. Melatonin vs. dexmedetomidine for sleep induction in children before electroencephalography. Front Pediatr. 2024 Apr 25;12:1362918. doi: 10.3389/fped.2024.1362918. eCollection 2024. PMID 38725985